CLINICAL TRIAL: NCT01961700
Title: In-hospital Physiotherapy for Patients Undergoing Thoracic Surgery - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Marcus Jonsson, Physiotherapist, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 122541
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Experimental): Physiotherapy (breathing exercises, mobilisation, exercises for upper limbs, advice on physical activity and exercise) provided daily during hospitalization.
  Interventions: Other: Physiotherapy
- Control group (No Intervention): No physiotherapy.

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy treatment
  Arms: Physiotherapy

SUMMARY:
Lung cancer is one of the most common types of cancer in the world, and the cancer that causes the most number of deaths. In Sweden, about 3700 persons are diagnosed every year. About one fifth of the patients are eligible for surgery.

Patients undergoing thoracic surgery suffer from pain and low health related quality of life after surgery.

In Australia, New Zealand, and the United Kingdom, pre- and postoperative physiotherapy is routinely provided for patients undergoing thoracic surgery, but the effects have not been thoroughly investigated. The scientific evidence of the effect of physiotherapy in connection with lung surgery is limited. The treatment typically consists of early mobilisation, breathing exercises and exercises for the shoulders. Reeve et al has shown that a postoperative shoulder exercise program can improve function and decrease pain after thoracotomy. Breathing exercises has not been found effective in reducing the rate of postoperative pulmonary complications after thoracic surgery.

The purpose of this study is to investigate the effect of in-hospital physiotherapy treatment, for patients undergoing thoracic surgery, on physical activity, health related quality of life, pain and lung function.

DETAILED DESCRIPTION:
Lung cancer is one of the most common types of cancer in the world, and the cancer that causes the most number of deaths. In Sweden, about 3700 persons are diagnosed every year. About one fifth of the patients are eligible for surgery.

Patients undergoing thoracic surgery suffer from pain and low health related quality of life after surgery.

In Australia, New Zealand, and the United Kingdom, pre- and postoperative physiotherapy is routinely provided for patients undergoing thoracic surgery, but the effects have not been thoroughly investigated. The scientific evidence of the effect of physiotherapy in connection with lung surgery is limited. The treatment typically consists of early mobilisation, breathing exercises and exercises for the shoulders. Reeve et al has shown that a postoperative shoulder exercise program can improve function and decrease pain after thoracotomy. Breathing exercises has not been found effective in reducing the rate of postoperative pulmonary complications after thoracic surgery.

The purpose of this study is to investigate the effect of in-hospital physiotherapy treatment, for patients undergoing thoracic surgery, on physical activity, health related quality of life, pain and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic surgery

Exclusion Criteria:

* Previous lung volume reducing surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-12; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Six minute walking test | up to 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Jonsson, PhD Student, Principal Investigator — Region Örebro län
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jonsson M, Hurtig-Wennlof A, Ahlsson A, Westerdahl E. Physical activity and health-related quality of life after lung cancer surgery- cross-sectional analyses 3 and 12 months postoperatively. Health Qual Life Outcomes. 2025 Jul 9;23(1):69. doi: 10.1186/s12955-025-02400-z. PMID 40629419
- [Derived] Jonsson M, Ahlsson A, Hurtig-Wennlof A, Vidlund M, Cao Y, Westerdahl E. In-Hospital Physiotherapy and Physical Recovery 3 Months After Lung Cancer Surgery: A Randomized Controlled Trial. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419876346. doi: 10.1177/1534735419876346. PMID 31530046
- [Derived] Jonsson M, Hurtig-Wennlof A, Ahlsson A, Vidlund M, Cao Y, Westerdahl E. In-hospital physiotherapy improves physical activity level after lung cancer surgery: a randomized controlled trial. Physiotherapy. 2019 Dec;105(4):434-441. doi: 10.1016/j.physio.2018.11.001. Epub 2018 Nov 20. PMID 30871894